CLINICAL TRIAL: NCT00896948
Title: Novel Protein Regulator of Tumor Suppressor ARF & NF-κB
Brief Title: Study of Proteins in Head and Neck Cancer Cells
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000558974; P30CA068485 (NIH); VU-VICC-HN-0529; VU-VICC-IRB-050259
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Head and Neck Cancer
Keywords: head and neck cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Blotting, Southern; Gene Expression Profiling; Flow Cytometry; Fluorescent Antibody Technique; Immunoenzyme Techniques; Immunohistochemistry; Immunologic Techniques

INTERVENTIONS:
Genetic: Southern blotting
Genetic: TdT-mediated dUTP nick end labeling assay
Genetic: gene expression analysis
Genetic: protein expression analysis
Other: flow cytometry
Other: fluorescent antibody technique
Other: immunoenzyme technique
Other: immunohistochemistry staining method
Other: immunologic technique

SUMMARY:
RATIONALE: Studying proteins in head and neck cancer cells in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This laboratory study is looking at proteins in head and neck cancer cells.

DETAILED DESCRIPTION:
OBJECTIVES:

* Define the function and mechanism of LZAP in regulating ARF.
* Determine the mechanism and biological consequences of LZAP inhibition of NF-κB.
* Determine if LZAP has tumor suppressor activity by conditional targeting of LZAP in mice.

OUTLINE: Using molecular laboratory techniques, this study examines the biochemical mechanisms by which LZAP activates transcriptional, tumor suppressive activity (both p53-dependent and p53-independent) of ARF and inhibits transcriptional, tumorigenic activity of NF-kB. LZAP regulation of newly identified ARF activities, such as S-phase delay and ARF-mediated B23 degradation are also evaluated. LZAP's tumor suppressive activity is assessed in vivo using a conditional knockout vector to target LZAP in mice and to observe for spontaneous and induced tumor formation. Laboratory analyses used to determine study endpoints include standard recombinant DNA, recombinant protein expression and purification, cell culture and transfection, cell labeling, reporter assays, flow cytometry, yeast-two hybrid, immunoprecipitation, immunoblotting, immunofluorescence, TUNEL assay, ELISA assay, Southern blotting, and protein and gene expression.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Head and neck cancer tumor cell line

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2005-05

PRIMARY OUTCOMES:
Function and mechanism of LZAP in regulating ARF
Mechanism and biological consequences of LZAP inhibition of NF-κB
Determination of LZAP tumor suppressor activity

CONTACTS AND LOCATIONS:
Overall Officials: Wendell G. Yarbrough, MD, FACS, Study Chair — Vanderbilt-Ingram Cancer Center
Locations (3):
- United States (3):
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Franklin, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee